CLINICAL TRIAL: NCT07010861
Title: Effects of Expressive Art Therapy Applied to Earthquake Victims Who Have Experienced Loss on Psychological Symptoms and Post-Traumatic Growth: A Randomized Controlled Study
Brief Title: Effects of Expressive Art Therapy Applied to Earthquake Victims Who Have Experienced Loss
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Kızılırmak Tatu (Other)
Responsible Party: Sponsor-Investigator, Merve Kızılırmak Tatu, Assisst. Prof. Dr., Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05.20.2024-E.950905
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Earthquake Victims
Keywords: Expressive Art Therapy; Earthquake Victims; Psychological Symptoms; Post-Traumatic Growth

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled intervention type study with a pre-test - post-test and follow-up, which is one of the quantitative research methods.
Who Masked: Participant
Masking Description: The study participants were assigned to the intervention and control groups using stratified block randomization. Block size and random assignment to the intervention and control groups were determined by an independent statistician. Participants in the study were stratified according to age (34 years and under, 35 years and over) and gender (female and male). Researcher blinding could not be performed because the researchers were involved in the implementation of the intervention program, data collection, and analysis phases. Participants were blinded by not disclosing which group they were in. In order to keep bias under control, the block group separation and randomization process of the stratified participants was performed by a statistician other than the researcher, and the researcher was not involved in this process. Data analysis was performed by an independent statistician who did not know the assignment and coding of the intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After the pre-test, the intervention program was started for the intervention group. The expressive arts therapy program was applied in six sessions, each session lasting 60-90 minutes. All sessions were conducted online. Each session started with greetings and mood control, then a brief evaluation of the previous week was made. The sessions consisted of three stages: giving instructions by the researcher, participants performing artistic actions with appropriate art elements and techniques, and participants working on sharing their artistic stimulation and associations. A list of materials to be used in the session (pencils, paint, paper, play dough, etc.) was sent to the participants one week before the sessions and they were asked to provide them until the session.
  Interventions: Other: Expressive Art Therapy
- Control (No Intervention): No intervention was made to the control group. After the follow-up test was applied to the participants in the experimental group, a three-session expressive arts therapy program was applied to the control group.

INTERVENTIONS:
Other: Expressive Art Therapy — As a strategy for coping with trauma, art production creates therapeutic effects on the individual with its sensory and physical aspects (Chapman, 2013; King-West and Hass-Cohen, 2008). When verbal expression is insufficient or carries the risk of re-traumatization, expressive art therapy offers a safe space through non-verbal expression (Talwar, 2007). It is stated that art production is effective in repairing self-integrity ruptures that occur in traumatic experiences (Harris, 2009). Through creative processes, the individual can restructure both internally and externally. Expressive art therapy, especially when applied in a group environment, creates a psychotherapeutic effect by providing participants with the opportunity to express their emotions, imagination and unconscious processes (Malchiodi, 2012; Kim et al., 2021). The commitment and reflective understanding that occur in group psychotherapy are among the factors that give hope and strength (Robb, 2017).
  Arms: Intervention

SUMMARY:
Earthquakes can negatively affect individuals' mental health by creating serious traumatic effects on individual and societal levels. Traumatic experiences such as losing one's home or workplace, being injured, or losing a loved one cause individuals to develop long-term psychological symptoms. In this context, strengthening psychosocial support programs aimed at coping with psychological and social problems after an earthquake is of great importance. In this study, the effect of expressive art therapy applied to individuals who experienced losses due to the earthquakes centered in Kahramanmaraş on psychological symptoms and post-traumatic growth was examined.

DETAILED DESCRIPTION:
A randomized controlled intervention design with pre-test-post-follow-up measurements was used, which is one of the quantitative research methods. In line with the power analysis, a total of 42 participants, 21 in each group, constituted the research sample. The distribution of participants to the intervention and control groups was made with stratified block randomization. The inclusion criteria of the study included being 18 years of age or older, knowing Turkish, and having experienced material and moral loss due to the earthquake; while the exclusion criteria were mental illness or receiving active psychosocial support. The Brief Symptom Inventory (BSI) and the Post-Traumatic Growth Scale (PTS) were used as data collection tools. The intervention process includes a six-session expressive arts therapy program. The scales will be administered online at pre-test, post-test and two-month follow-up. Data will be evaluated with repeated measures and two-way variance analyses. It is expected that this study will contribute to post-traumatic recovery processes and art-based psychosocial interventions.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Being able to understand, speak and write Turkish,
* Having directly experienced the earthquakes centered in Kahramanmaraş, -
* Having experienced material and moral losses due to the earthquakes centered in Kahramanmaraş

Exclusion Criteria:

* Having a neurological disorder that prevents communication,
* Actively receiving any psychosocial support/counseling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Brief Symptom Inventory (BSI) | Change from baseline to 6 weeks (also assessed at 14 weeks post-baseline)
  It is a 53-item symptom screening scale developed by Derogatis. The scale consists of 9 subscales and 3 global indexes. The 9 subscales of the scale are, respectively, Somatization (S) (items 2, 7, 23, 29, 30, 33, 37), Obsessive-compulsive disorder (OCD) (items 5, 15, 26, 27, 32, 36), Interpersonal sensitivity (IS) (items 20, 21, 22, 42), Depression (D) (items 9, 16, 17, 18, 35, 50), Anxiety disorder (AD) (items 1, 12, 19, 38, 45, 49), Hostility (H) (items 6, 13, 40, 41, 46), Phobic anxiety (PA) (items 8, 28, 31, 43, 47), Paranoid ideation (PD) (items 4, 10, 24, 48, 51) and Psychoticism (P) (items 3, 14, 34, 44, 53). Additional items (EM) (items 11, 25, 39, 52) include items related to eating and drinking disorders, sleep disorders, death and thoughts about death, and feelings of guilt. The global indices are the Disorder Severity Index, the Symptom Total Index, and the Symptom Disorder Index, respectively.
Post-Traumatic Growth Scale (PTGS) | Change from baseline to 6 weeks (also assessed at 14 weeks post-baseline)
  The Posttraumatic Growth Inventory was developed by Tedeschi and Calhoun (1996) to measure the development that occurs in individuals after trauma. The scale consists of 21 items and the items are scored on a 6-point scale from 0 to 5. The scores obtained from the scale vary between 0 and 105, and a high score indicates that the person has experienced a positive change, that is, growth, after the trauma. Factor analysis determined that the scale has 5 sub-dimensions (positive change in interpersonal relationships, awareness of new opportunities, understanding the value of life, increasing personal resilience, and strengthening spirituality). The internal consistency coefficient of the scale was reported as .93 (Kağan et al., 2012).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, ÇANKAYA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Other researchers wiil be able to read detailed information such as the research method and results when the research is published. The "Research Protocol" will be available on this PRS page.